CLINICAL TRIAL: NCT01203020
Title: Once Daily Intravenous Busulfex as Part of Reduced-toxicity Conditioning for Patients With Relapsed/Refractory Hodgkin's and Non-Hodgkin's Lymphomas Undergoing Allogeneic Hematopoietic Progenitor Cell Transplantation - A Multicenter Phase II Study
Brief Title: Once Daily Targeted Intravenous (IV) Busulfex as Part of Reduced-toxicity Conditioning for Patients With Refractory Lymphomas Undergoing Allogeneic Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVU 11310
Record Dates: First submitted 2010-09-13; First posted 2010-09-16 (Estimated); Results first posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Hodgkin's; non-Hodgkin's; lymphomas; allogeneic hematopoietic progenitor cell transplant; HPCT; busulfex; fludarabine; reduced-toxicity conditioning; reduced-intensity conditioning
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma | interventions — Busulfan; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic hematopoietic progenitor cell transplant (Experimental): Intravenous busulfex 130mg/m2 on days -6 to -3 before transplant
  Interventions: Drug: Busulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Busulfan — Busulfex 130 mg/m2 intravenous piggy back (IVPB) for 4 days (Day -6 to -3) pharmacokinetic (PK) samples for Busulfex dose adjustment drawn on Day -6
  Other Names: Busulfex
Drug: Fludarabine — Fludarabine 40 mg/m2 IVPB for 4 days (Day -6 to -3)
  Other Names: Fludarabine Monophosphate; Fludara

SUMMARY:
This is a phase II study of allogeneic hematopoietic progenitor cell transplantation (HPCT) followed reduced toxicity conditioning with once daily intravenous Busulfex and fludarabine in patients with relapsed/chemotherapy refractory Hodgkin's and non-Hodgkin's lymphomas.

DETAILED DESCRIPTION:
This study hopes to learn if giving intravenous (IV) busulfan with fludarabine before (as a conditioning regimen) allogeneic hematopoietic progenitor cell transplantation (HPC) is safe and helps patients with Non-Hodgkin´s Lymphoma (NHL) and Hodgkin´s Lymphoma (HL). An HPC transplant takes cells from a donor´s bone marrow and, after chemotherapy treatment with a conditioning regimen, infuses the donor´s cells into the patient´s body. Busulfan is a strong drug that suppresses the immune system and fludarabine is a chemotherapy (cancer fighting) drug. These drugs can stop the growth of cancer cells by breaking the Deoxyribonucleic acid (DNA) or genetic material which is necessary for the growth of both healthy and cancer cells. The use of IV busulfan with fludarabine as a conditioning regimen prior to HPC transplant is investigational (not approved by the Food and Drug Administration [FDA]).

Busulfan is only given once daily by IV in this study, which is also not approved by the FDA. Patients in this study will go through standard procedures for their disease like medical history, physical exam, blood tests, Multi Gated Acquisition Scan (MUGA) scan or echocardiogram, bone marrow aspirate or biopsy, and lung functions test. Patients will be asked to donate additional blood and bone marrow for this study and for potential future research on their blood related to this study. Because of the normal procedures for HPC transplants patients in this study will be hospitalized for 4 to 6 weeks or longer and will make frequent trips to the clinic to visit the study doctor for supervision for at least one year. Each patient will also have to have a central venous catheter inserted into a large vein above the heart. This is used to give the drugs and to take blood samples.

Participation in this study will last about two years. The study expects to enroll 32 patients and will open to at least two collaborating institutions in the future. Upon initial Institutional Review Board (IRB) approval enrollment will only occur at West Virginia University (WVU). The IRB will be notified before enrollment occurs at other institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years of age are eligible.
2. Eligible histologies include:

   * B-cell, T-cell or NK-cell NHL refractory to frontline or salvage therapy defined as failure to achieve complete or partial remission according to standard criteria.
   * Diffuse large B-cell lymphoma relapsing within 12 months of finishing a rituximab containing first line chemotherapy regimen (regardless of response to salvage chemotherapy)or with evidence of c-myc. Primary refractory NHL (regardless of response to salvage chemotherapy).
   * Hodgkin lymphoma which is chemorefractory after at least two prior therapies.
   * Hodgkin and NHL in an untreated relapse.
   * Transformed NHL or chronic lymphocytic leukemia undergoing Richter's transformation (regardless of response to last chemotherapy). Patients with chemosensitive relapsed NHLs or Hodgkin lymphoma, but considered ineligible for curative therapy with autologous transplantation, because of (a) inability to collect stem cells, (b) prior autografting, (c) presence of myelodysplasia or (d) histology not considered curable with autografting in opinion of treating physician will be eligible.
3. All patients must have at least one suitable HLA-matched sibling or volunteer unrelated donor available (according to institutional guidelines). HLA typing should be performed at least at serological level for HLA-A, -B, and -C and at allele level for HLA-DRB1. One antigen or allele level mismatch will be permitted between the donor and the recipient; however each donor/recipient pair must match at HLA-DRB1 at allele level.
4. Patient must be able to provide informed consent.
5. Left ventricular ejection fraction ≥ 40%. No uncontrolled arrhythmias or uncontrolled New York Heart Association class III-IV heart failure.
6. Bilirubin, aspartate aminotransferase (AST), and Alanine transaminase (ALT) ≤ 3 x normal; and absence of hepatic cirrhosis.
7. Adequate renal function as defined by a serum creatinine clearance of ≥ 40% of normal calculated by Cockcroft-Gault equation.
8. DLCO (diffusion capacity; corrected for hemoglobin) or forced expiratory volume (FEV1) ≥ 50% of predicted.
9. Karnofsky performance status ≥ 70.
10. A negative pregnancy test will be required for all women of child bearing potential. Breast feeding is not permitted.

Exclusion Criteria:

1. Patients eligible for potentially curative therapy with autologous transplantation.
2. Patients with lymphoblastic lymphoma.
3. Patients with positive human immunodeficiency virus (HIV) serology.
4. Clinical evidence of uncontrolled bacterial, viral or fungal infection at the time of transplant conditioning.
5. Prior allogeneic transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10-12 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Kanate, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 53.50 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of 1 Year Overall Survival (OS)
Description: Percentage of participants--1 year overall survival (OS) following transplantation.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
percentage of participants | 63.6 [46.4 to 87.3]

2. Primary Outcome: Percentage of 2 Year Overall Survival (OS)
Description: Percentage of participants-- 2 Year Overall Survival (OS) post transplant
Time Frame: At 2nd year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
percentage of participants | 59.1 [41.7 to 83.7]

3. Primary Outcome: Percentage of 1-year Progression Free Survival (PFS)
Description: Percentage of 1-year progression free survival (PFS) of patients with chemotherapy refractory Hodgkin's and non-Hodgkin's lymphoma (NHL) undergoing reduced-toxicity conditioning (RTC) with once daily intravenous Busulfex and fludarabine.
Time Frame: At 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
percentage of participants | 59.1 [41.7 to 83.7]

4. Primary Outcome: Percentage of 2-year Progression Free Survival (PFS)
Description: Percentage of 2-year progression free survival (PFS) of patients with chemotherapy refractory Hodgkin's and non-Hodgkin's lymphoma (NHL) undergoing reduced-toxicity conditioning (RTC) with once daily intravenous Busulfex and fludarabine.
Time Frame: At 2 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
percentage of participants | 45.5 [28.8 to 71.8]

5. Secondary Outcome: Relapse Rate (RR) Following Transplantation at 1-year.
Description: Percentage of participants Relapse Rates (RR) following transplantation at 1-year.
Time Frame: At 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
percentage of participants | 28.7 [6.3 to 45.8]

6. Secondary Outcome: Relapse Rate (RR) Following Transplantation at 2-year.
Description: Percentage of participants Relapse Rates (RR) following transplantation at 2-year.
Time Frame: At 2 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
percentage of participants | 39.7 [13.7 to 57.9]

7. Secondary Outcome: Non-Relapse Mortality (NRM) Following RTC Transplantation at 1 Year.
Description: Percentage of participants NRM following RTC transplantation at 1-year.
Time Frame: At 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
percentage of participants | 17.1 [0.0 to 33.1]

8. Secondary Outcome: Non-Relapse Mortality (NRM) Following RTC Transplantation at 2 Years.
Description: Percentage of participants NRM following RTC transplantation at 2-year.
Time Frame: At 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
percentage of participants | 24.6

9. Secondary Outcome: Rates of Acute and Chronic Graft Versus Host Disease (GVHD).
Description: Count/Percentage rates of acute and chronic graft versus host disease (GVHD).
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
Number analyzed (Participants) | 22
Participants
  Acute GVHD | 5
  Chronic GVHD | 3

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Allogeneic Hematopoietic Progenitor Cell Transplant
All-Cause Mortality (participants affected / at risk) | 9/22
Serious Adverse Events (participants affected / at risk) | 9/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Hematopoietic Progenitor Cell Transplant (N=22)
Death (General disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-10-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT01203020/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT01203020/ICF_001.pdf